CLINICAL TRIAL: NCT06592027
Title: Optimal Dose of Dexmedetomidine for Attenuation of Endotracheal Intubation Pressor Response Using Cardiometry. a Randomized, Double-blinded Study
Brief Title: Dexmedetomidine for Attenuation of Pressor Response
Acronym: Precedex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Moshira sayed mohamed, Lecturer of anesthesia and intensive care, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT (811)
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pressor Response
Keywords: Dexmedetomidine; pressor response; optimum dose

STUDY DESIGN:
Intervention Model Description: The aim of our study is to assess and compare the efficacy of two different doses of dexmedetomidine (0.5 μg/kg and 1.0 μg/ kg) to find out its optimal dose in attenuation of hemodynamic pressor response to laryngoscopy and intubation with the use of Cardiometry for continuous CO monitoring beat by beat.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Placebo Comparator): this group will receive single dose of dexmedetomidine 0.5 mcg /kg in 50 ml normal saline over 10 min IV infusion
  Interventions: Drug: PRECEDEX INJ★ 2ML
- Group B (Active Comparator): this group will receive single dose of dexmedetomidine 1 mcg /kg in 50 ml normal saline over 10 min IV infusion
  Interventions: Drug: PRECEDEX INJ★ 2ML

INTERVENTIONS:
Drug: PRECEDEX INJ★ 2ML — this group will receive single dose of dexmedetomidine 0.5 mcg /kg in 50 ml normal saline over 10 min IV infusion
  Arms: Group A
Drug: PRECEDEX INJ★ 2ML — single dose of dexmedetomidine 1 mcg /kg in 50 ml normal saline over 10 min IV infusion
  Arms: Group B

SUMMARY:
Direct laryngoscopy and tracheal intubation are usually associated by hemodynamic changes due to increased sympathoadrenal activity which could precipitate serious negative effects in compromised patients . The pressor response could be blunted by dexmedetomidine which is a selective alpha 2 agonist which might provide hemodynamic stability during tracheal intubation.

DETAILED DESCRIPTION:
Various drugs include local anesthetics, beta-blockers, calcium channel blockers, and narcotic analgesics have been tried to blunt the laryngoscopy and intubation response, with varied success. Dexmedetomidine is a potent and highly selective alpha-2 receptor agonist with sympatholytic, sedative, amnestic, and analgesic properties. Its various effects have led to its increasing use for reducing anesthetic and analgesic requirements in the perioperative period. It inhibits sympathetic activity thus terminating the pain signals and thereby blunts the pressor response associated with laryngoscopy and endotracheal intubation. Electrical cardiometry is recently introduced for assessment of many cardiovascular variables and continuously applicable method of cardiac output (CO), stroke volume (SV), and other hemodynamic parameters monitoring. Its use is growing because it is non-invasive, shows reliability in CO measurements and can be used as a continuous bedside monitor Although different doses of dexmedetomidine (0.5- 2.0 μg/kg) have been used in various studies which suggested its efficacy in blunting the hemodynamic pressor response , However, no studies to the best of our knowledge had incorporated CO monitoring for detection of minimal hemodynamic changes during laryngoscopy and endotracheal intubation which can be best achieved by using Cardiometry monitor.

In this study, we will compare two doses of dexmedetomidine for prophylaxis against pressor response of ETI using cardiometry.

ELIGIBILITY:
Inclusion Criteria:

1 - ASA physical status 1-2. 2. Age 18- 60 years old of both sexes. 3. Patients undergoing elective surgery under general anesthesia and tracheal intubation.

Exclusion Criteria:

1. Age < 18 years and ≥ 60 years
2. Pregnancy
3. Emergency surgery or full stomach
4. Renal or Hepatic patients
5. Patients with suspected difficult airway {e.g., high neck circumference, high body mass index (above 30 kg/m2), airway masses, mouth scars, neck scars, limited neck extension or history of snoring.
6. Total duration of laryngoscopy will be noted and in cases where duration exceeded 15 sec the case will be excluded from the study.
7. Any patient on regular intake of beta blockers or calcium channel blockers
8. Patients with any known hypersensitivity or contraindication to dexmedetomidine,
9. Patients with significant neurological, psychiatric, or neuromuscular disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Heart rate measurment | after 1 minute of successful tracheal intubation
  single measurement after intubation

SECONDARY OUTCOMES:
cardiac output | from the start of induction of anesthesia till 5 minutes after successful tracheal intubation
  serial measurements every 1 minute

CONTACTS AND LOCATIONS:
Overall Officials: Moshira Sayed Lecturer of anesthesia and intensive care, M.D., Principal Investigator — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz Research institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will be available upon request from the principal investigator

REFERENCES:
- [Background] Misra S, Behera BK, Mitra JK, Sahoo AK, Jena SS, Srinivasan A. Effect of preoperative dexmedetomidine nebulization on the hemodynamic response to laryngoscopy and intubation: a randomized control trial. Korean J Anesthesiol. 2021 Apr;74(2):150-157. doi: 10.4097/kja.20153. Epub 2020 May 20. PMID 32434291